CLINICAL TRIAL: NCT03213249
Title: Bacterial Biofilms in Reconstructive Breast Prostheses Following Mastectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Plastic Surgery Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 201704134
Record Dates: First submitted 2017-06-22; First posted 2017-07-11 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Breast Implant Infection; Mammoplasty
MeSH Terms: interventions — Saline Solution; Cefazolin; Tissue Expansion Devices; Breast Implants; Gentamicins; Bacitracin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Intraoperative pocket irrigation with NS (Active Comparator): * 1 gram cefazolin intravenous before surgical incision
  * Standard of care bilateral skin- or nipple-sparing mastectomies as determined by breast surgical oncologists
  * Immediate standard of care breast reconstruction with subpectoral tissue expanders and a 16 x 8 ADM sling
  * Standard of care saline pocket irrigation will receive 500 cc of normal saline alone per pocket.
  Interventions: Other: Normal saline; Procedure: Skin biopsy; Procedure: Bilateral skin- or nipple-sparing mastectomies; Device: Tissue expander; Device: Breast implant; Procedure: Autologous flap; Other: Acellular dermal matrix sling
- Arm 2: Intraoperative pocket irrigation with NS + antibiotics (Active Comparator): * 1 gram cefazolin intravenous before surgical incision
  * Standard of care bilateral skin- or nipple-sparing mastectomies as determined by breast surgical oncologists
  * Immediate standard of care breast reconstruction with subpectoral tissue expanders and a 16 x 8 ADM sling
  * Standard of care antibiotic pocket irrigation will receive 500 cc of normal saline plus 1 gram cefazolin, 80 mg gentamicin, and 50,000 units bacitracin
  Interventions: Other: Normal saline; Drug: Cefazolin; Procedure: Skin biopsy; Procedure: Bilateral skin- or nipple-sparing mastectomies; Device: Tissue expander; Device: Breast implant; Procedure: Autologous flap; Other: Acellular dermal matrix sling; Drug: Gentamicin; Drug: Bacitracin

INTERVENTIONS:
Other: Normal saline — Intraoperative pocket irrigation with normal saline
  Other Names: NS
Drug: Cefazolin — Cefazolin, gentamicin, and bacitracin will be mixed together in 1 L of normal saline and placed in the pocket created by the breast once it is removed
  Other Names: Ancef
  Arms: Arm 2: Intraoperative pocket irrigation with NS + antibiotics
Procedure: Skin biopsy — Biopsies will be taken from the skin at the time of mastectomy and at the time of implant exchange.
Procedure: Bilateral skin- or nipple-sparing mastectomies — Standard of care
Device: Tissue expander — Standard of care
Device: Breast implant — * Standard of care
  * Either breast implant or autologous flap
Procedure: Autologous flap — * Standard of care
  * Either breast implant or autologous flap
Other: Acellular dermal matrix sling — Standard of care
Drug: Gentamicin — Cefazolin, gentamicin, and bacitracin will be mixed together in 1 L of normal saline and placed in the pocket created by the breast once it is removed
  Other Names: Garamycin
  Arms: Arm 2: Intraoperative pocket irrigation with NS + antibiotics
Drug: Bacitracin — Cefazolin, gentamicin, and bacitracin will be mixed together in 1 L of normal saline and placed in the pocket created by the breast once it is removed
  Arms: Arm 2: Intraoperative pocket irrigation with NS + antibiotics

SUMMARY:
Breast implants, either cosmetic or reconstructive, are among the most common procedures performed by plastic surgeons. Bacterial infections or biofilms are implicated in the majority of breast implant complications including infection requiring explantation, capsular contracture (CC), and/or breast-implant associated anaplastic large cell lymphoma (BIA-ALCL). The research team, which has already extensively characterized bacterial pathogenesis in the urinary tract and designed non-antibiotic therapeutics to reduce the incidence of catheter-associated urinary tract infections (CAUTIs), and proposal will study bacteria-breast implant interactions and explore further the impact of the breast microbiome. The proposed research provides a greater understanding of which bacteria can colonize breast implants, their source, and how effective antibiotic pocket irrigation is at eliminating them, and begins to examine the mechanisms by which bacteria bind and colonize the implant surface. These insights will set the groundwork for developing new therapeutic agents that can disrupt the binding of certain bacteria to breast implants. Strategies that minimize problems bacteria can cause, while avoiding antibiotics, will reduce bacteria-related implant complications, limit antibiotic-related side effects, and reduce bacterial resistance.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Between 18 and 75 years of age, inclusive
* Undergoing bilateral mastectomy reconstruction with tissue expanders (ipsilateral therapeutic/contralateral prophylactic) planned to be exchanged for breast implants
* Able to understand and willing to sign an IRB-approved written informed consent document

Exclusion Criteria:

* Male

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
Number of tissue expander(s) removed due to infection | Up to 1 year
  The bulk of analyses will be to study bacterial biofilm formation on the explanted breast tissue, skin/scar, drain, acellular dermal matrix, tissue expander, and capsule.
Number of tissue expander(s) removed due to patient preference | Up to 1 year

SECONDARY OUTCOMES:
Duration of implantation | Up to 1 year
Duration the drain was in | Up to 1 year
Incidence of development of an infection or a wound | Up to 1 year
Incidence of capsular contracture | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Terence M Myckatyn, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu